CLINICAL TRIAL: NCT06396078
Title: Improvement of PPROM Management With Prophylactic Antimicrobial Therapy
Brief Title: Improvement of PPROM Management With Prophylactic Antimicrobial Therapy (iPROMPT)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Kartik K Venkatesh, Principal Investigator, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024H0122
Record Dates: First submitted 2024-04-25; First posted 2024-05-02 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Preterm Premature Rupture of Membrane; Pregnancy, High Risk; Preterm Birth
Keywords: Pregnancy; Preterm premature rupture of membranes; Latency; Chorioamnionitis; Antibiotic prophylaxis
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes; Premature Birth; Chorioamnionitis | interventions — Ceftriaxone; Clarithromycin; Metronidazole; Amoxicillin; Azithromycin; Erythromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Participants randomized to the intervention group will receive the following regimen:
  * Ceftriaxone 1 g IV q 24 hours x 7 days
  * Clarithromycin 500 mg PO BID x 7 days
  * Metronidazole 500 mg PO q 12 hours x 7 days
  Interventions: Drug: Ceftriaxone 1000 MG; Drug: Clarithromycin 500mg; Drug: Metronidazole 500 mg
- Standard of care (Other): Participants randomized to the standard care group will receive the following regimen:
  * Ampicillin 2 g IV q 6 hours x 48 hours followed by amoxicillin 250 mg q 8 hours for an additional 5 days
  * Azithromycin 1 g PO x 1 dose OR erythromycin 250 mg IV q 6 hours x 48 hours followed by erythromycin 333 mg PO TID for an additional 5 days
  Interventions: Drug: Ampicillin 2 GM Injection; Drug: Amoxicillin 250 MG; Drug: Azithromycin; Drug: Erythromycin

INTERVENTIONS:
Drug: Ceftriaxone 1000 MG — Ceftriaxone 1 g IV q 24 hours x 7 days (in addition to clarithromycin and metronidazole)
  Arms: Intervention group
Drug: Clarithromycin 500mg — Clarithromycin 500 mg PO BID x 7 days (in addition to ceftriaxone and metronidazole)
  Arms: Intervention group
Drug: Metronidazole 500 mg — Metronidazole 500 mg PO q 12 hours x 7 days (in addition to clarithromycin and ceftriaxone)
  Arms: Intervention group
Drug: Ampicillin 2 GM Injection — Ampicillin 2 g IV q 6 hours x 48 hours (prior to amoxicillin and in addition to either azithromycin or erythromycin)
  Arms: Standard of care
Drug: Amoxicillin 250 MG — Amoxicillin 250 mg q 8 hours for an additional 5 days (following ampicillin and in addition to either azithromycin or erythromycin)
  Arms: Standard of care
Drug: Azithromycin — Azithromycin 1 g PO x 1 dose (in addition to ampicillin and amoxicillin)
  Arms: Standard of care
Drug: Erythromycin — Erythromycin 250 mg IV q 6 hours x 48 hours followed by erythromycin 333 mg PO TID for an additional 5 days (in addition to ampicillin and amoxicillin)
  Arms: Standard of care

SUMMARY:
To conduct an unblinded pragmatic randomized controlled trial (pRCT) "Improvement of PPROM Management with Prophylactic Antimicrobial Therapy (iPROMPT)" of a seven-day course of ceftriaxone, clarithromycin, and metronidazole versus the current standard of care of a seven-day course of ampicillin/amoxicillin and azithromycin or erythromycin to prolong pregnancy and decrease adverse perinatal outcomes among hospitalized pregnant individuals undergoing expectant management of PPROM <34 weeks.

DETAILED DESCRIPTION:
Preterm prelabor rupture of membranes (PPROM) is the most common identifiable risk factor associated with preterm birth and affects 1 in 3 pregnant individuals in the United States with spontaneous preterm birth. Individuals diagnosed with PPROM who meet criteria for expectant management are currently admitted to the hospital for observation until delivery, which is generally recommended at 34 weeks' gestation unless indicated sooner. Initially upon admission, a course of prophylactic antibiotics is administered as this has been shown to prolong pregnancy and improve neonatal outcomes. The standard antibiotic regimen, primarily based on data published in 1997, includes ampicillin followed by amoxicillin with erythromycin or azithromycin for a total of 7 days. Ongoing studies are needed to determine the optimal prophylactic antibiotic regimen given changes in bacterial sensitivities over time, lack of adequate coverage for common organisms including genital mycoplasma, inadequate placental transfer of currently used antibiotic agents, ineffective antibiotic response at reducing the fetal inflammatory response, and new promising antibiotic agents that address these limitations. A promising expanded-spectrum alternative regimen with proof-of-concept is ceftriaxone, clarithromycin, and metronidazole. Observational studies have shown successful eradication of intraamniotic inflammation/infection using this new regimen. This regimen offers multiple potential advantages, including: higher bioavailability, higher transplacental transfer, and effectiveness against genital mycoplasma (clarithromycin), greater anaerobic coverage (metronidazole), and a longer half-life and expanded coverage against gram-negative bacteria (ceftriaxone) compared with the current standard regimen.

ELIGIBILITY:
Inclusion criteria

* Admitted to the inpatient unit for expectant management of PPROM until delivery
* Age ≥ 18 years with the ability to provide informed consent
* Gestational age between 23 0/7 and 32 6/7 weeks

Exclusion criteria

* Having received more than one dose of any prophylactic antibiotic
* Suspected or confirmed infection requiring treatment with antibiotics
* Allergy or contraindication to an antibiotic in either arm
* Maternal immunosuppression

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is restricted to pregnant individuals.
Enrollment: 56 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Latency | From randomization to delivery
  Latency will be measured in hours, and also reported as days for clinical interpretability.

SECONDARY OUTCOMES:
Neonatal outcome composite checklist | From birth to up to 6 weeks postpartum
  Includes neonatal sepsis, respiratory distress syndrome, any mechanical ventilation, bronchopulmonary dysplasia, intraventricular hemorrhage, periventricular leukomalacia, necrotizing enterocolitis, stillbirth, or neonatal death
Endometritis | From birth to up to 6 weeks postpartum
  Diagnosed If the patient develops two of the following 1) oral body temperature ≥101°F at any time, or a temperature of ≥100.4 °F 24 hours after delivery, 2) maternal tachycardia that parallels the temperature, 3) uterine tenderness, 4) purulent vaginal discharge, or 5) associated findings with advanced endometritis (dynamic ileus, pelvic peritonitis, pelvic abscess, bowel obstruction, necrosis of the lower uterine segment)
Surgical site infection | From birth to up to 6 weeks postpartum
  Presence of either superficial or deep incisional SSI described as cellulitis/erythema and induration around the incision or purulent discharge from the incision site, with or without fever, such as necrotizing fasciitis (diagnosed based on necrotizing wound infection). Intraabdominal abscess may or may not be present. Wound hematoma, seroma, or incisional breakdown alone in the absence of the above signs does not constitute infection.
Individual clinical infections | From birth to up to 6 weeks postpartum
Puerperal fever | From birth to up to 6 weeks postpartum
  temperature ≥ 100.4 °F at least twice 30 minutes apart, or once with the use of antipyretic, or ≥ 101 °F once. This will be analyzed for intrapartum and postpartum fever.
Histopathologic chorioamnionitis/funisitis on histologic placental evaluation | From randomization to delivery
Antibiotic receipt postpartum | From birth to up to 6 weeks postpartum
Adverse events | From randomization to delivery
  Allergic reactions (anaphylaxis, angioedema, urticaria), Stevens Johnsons syndrome, gastrointestinal side effects (nausea, vomiting, constipation, diarrhea, ileus)

CONTACTS AND LOCATIONS:
Overall Officials: Marissa Berry, MD, Principal Investigator — Ohio State University; Kartik K Venkatesh, MD, PhD, Principal Investigator — Ohio State University
Locations (2):
- United States (2):
  - The Ohio State University Wexner Medical Center OB/GYN Maternal and Fetal Medicine, Columbus, Ohio
  - University of Texas Medical Branch, Galveston, Texas

IPD SHARING:
Plan to Share IPD: No